CLINICAL TRIAL: NCT01458470
Title: A Trial of Memantine as Symptomatic Treatment for Early Huntington Disease; a Phase IIb Study
Brief Title: A Trial of Memantine as Symptomatic Treatment for Early Huntington Disease
Acronym: MITIGATE-HD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Huntington Society of Canada (Other); Huntington Study Group (Network)
Responsible Party: Principal Investigator, Blair Leavitt, Associate Professor, Department of Medical Genetics, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H11-01364
Record Dates: First submitted 2011-10-20; First posted 2011-10-24 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Huntington Disease
Keywords: huntington; huntingtin; memantine; ebixa; namenda
MeSH Terms: conditions — Huntington Disease | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Memantine (Active Comparator): NMDA Receptor Antagonist
  Interventions: Drug: Memantine
- Sugar pill (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Memantine — oral tablet, 1 BID, 24 weeks
  Other Names: Ebixa; DIN 02260638; Namenda
  Arms: Memantine
Other: Placebo — oral tablet, 1 BID, 24 weeks
  Arms: Sugar pill

SUMMARY:
Huntington disease is characterized by difficulties in movement and thinking. Psychological disturbances including irritability, aggression, loss of interest, depressed mood, obsessions and compulsions, also represent common symptoms of HD. These symptoms are distressing both for HD patients and their caregivers, contribute to the loss of ability to carry out activities of daily living, and present a major treatment challenge for physicians. The goal of this study is to determine the effect of memantine on movement, thinking and emotional difficulties in HD patients. Memantine is a medication originally approved for the treatment of aggression and agitation in patients with moderate-to-severe Alzheimer's disease (AD), which has also recently been shown to improve the behavioural and neuropathological symptoms in a mouse model of Huntington Disease (HD).

DETAILED DESCRIPTION:
TRACK-HD was a multi-centre, multi-national, prospective, observational study of pre-manifest and early Huntington's disease (HD) with a control group of volunteers not carrying the HD mutation. The goal of the project was to contribute essential methodology that will form the basis for clinical trials in pre-manifest and early HD. TRACK-HD complemented existing observational studies (e.g., Predict-HD, PHAROS, COHORT), sharing some features, but also having areas of unique emphasis.

The UBC site recruited 90 subjects including 30 control subjects, 30 asymptomatic pre-manifest HD gene carriers and 30 subjects with early symptoms of HD (stage 1 or 2). All subjects were assessed using the TRACK-HD battery at baseline, 1 year, 2 years, and 3 years. Following the fourth visit (3 year assessment), the TRACK-HD study will be completed, and the 30 subjects with early symptoms of HD will be invited to enroll in the MITIGATE-HD Study.

The MITIGATE-HD study is a single center Phase IIb,out-patient,randomized, double-blind, placebo-controlled trial of memantine treatment in subjects with Huntington disease (HD). The study will evaluate Memantine 10 mg two times daily (BID) administered orally (PO) for six months (24 weeks) compared with matching placebo BID. Safety and tolerability will be assessed by recording of adverse events and by monitoring of vital signs, physical examinations, and suicidality risk scores.

The TRACK-HD assessment battery will be administered to all subjects after six months of study drug administration. The effects of memantine will be evaluated both against placebo as well as compared to the previous 3 years of observational data from the TRACK-HD Study.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the study, a subject must be enrolled in the early HD cohort of the TRACK-HD study and:

* be at least 18 years of age and not older than 65
* able to provide written consent
* carry the abnormal HD gene and show early symptoms of HD
* be able and willing to comply with study requirements, including travel to study center
* have no metal implants to be suitable for MRI scans and able to tolerate them
* able to tolerate blood draws
* be of stable medical, psychiatric and neurological health at the time of enrollment
* not have a history of significant head injury
* not have a history of significant hand injury that would prevent either writing or performing rapid computer tasks
* not be abusing drugs and/or alcohol that may cause failure to comply with study procedures
* not be currently participating in PREDICT-HD or a clinical drug trial.

Exclusion Criteria:

Prospective subjects will be excluded if:

* they are younger than 18 years of age and older than 65
* they are unable to provide written consent
* they show advanced symptoms of HD if they are HD gene carriers
* they are unwilling to comply with study requirements, including travel to study center
* they are unsuitable for MRI (e.g, claustrophobia, metal implants) or unable to tolerate them
* they are unable to tolerate blood draws; or,
* they have a major psychiatric disorder, concomitant significant neurological disorder or concomitant significant medical illness at the time of enrollment
* they have a history of CNS disease or significant head injury; or,
* they have a history of significant hand injury that would prevent either writing or performing rapid computer tasks; or,
* they are likely to be non-compliant with study procedures due to drug and/or alcohol abuse; or,
* they are participating in PREDICT-HD or a clinical drug trial at the time of enrollment.
* they are not sighted
* English is not their first language
* they are currently or treated within the last 6 months with antipsychotic medications, including the traditional neuroleptics such as haloperidol as well as the atypical antipsychotics risperidone, clozapine, quetiapine and olanzapine
* they are use phenothiazine-derivative antiemetic medications such as prochlorperazine, metoclopramide, promethazine and Inapsine on a regular basis (greater than 3 times per month)
* they have a history of learning disability and/or mental retardation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-09; Primary Completion 2012-08 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Utility of TRACK-HD study endpoints in a clinical trial setting | 24 weeks
  To examine the clinical utility of novel trial endpoints (such as Putaminal NAA measured by MRS) developed in the TRACK-HD study in the setting of a placebo-controlled therapeutic trial.

SECONDARY OUTCOMES:
Neuropsychiatric and Cognitive Test Scores | 24 weeks
  To examine effect of memantine versus placebo on the scores of: a) the irritability and agitation/aggression sub-categories of the Neuropsychiatric Inventory (NPI), and also the total NPI, b) cognitive tests: Circle Tracing , Symbol Digit Modality, Stroop Word Reading, and Spot the Change, c) total HD-ADL, d) total UHDRS, and the UHDRS sub-scale: Cognitive, Behavioural, Functional, and Independence scales. e) In patients recruited at the UBC study site, the effect on striatal N-acetyl aspartate levels (a measure of neuronal dysfunction) will be assessed by Magnetic Resonance Spectroscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Blair R. Leavitt, MD,CM,FRCPC, Principal Investigator — University of British Columbia; Michael R. Hayden, MD,ChB,PhD, Study Chair — The University of British Columbia
Locations (1):
- The Centre for Huntington Disease, Vancouver, British Columbia, Canada

REFERENCES:
- See also: The Huntington Study Group — http://www.huntington-study-group.org/
- See also: The Huntington Society of Canada — http://www.huntingtonsociety.ca/
- See also: Health Canada — http://www.hc-sc.gc.ca